CLINICAL TRIAL: NCT06866639
Title: Cognitive Behavioural Therapy/Metacognitive Therapy for Low Self Esteem
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Roger Hagen, Professor, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSE06064685
Record Dates: First submitted 2025-02-13; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Psychological Disorders
Keywords: low self esteem; cognitive behavioural therapy; metacognitive therapy; depressive symptoms; anxiety symptoms
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The first group (n=10) will be treated with MCT, whereas the second group (n = 10) will be treated with CBT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): Cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy
- Metacognitive therapy (Experimental): Metacognitive therapy
  Interventions: Behavioral: Metacognitive therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The CBT is based on the treatment manual written by Fennell (1997). The patients receiving CBT will be treated for 8 sessions, with weekly session of 45-60 minutes duration.
  Arms: Cognitive behavioral therapy
Behavioral: Metacognitive therapy — The meta-cognitive treatment program is based on Wells's metacognitive therapy (Wells, 2013). The patients receiving meta-cognitive therapy will be treated for 8 sessions, with weekly session of 45-60 minutes duration.
  Arms: Metacognitive therapy

SUMMARY:
The goal for this clinical trial is to explore the effect of CBT/MCT on the treatment of low self esteem. 20 patients with low self-esteem will be selected and distributed into two either MCT or a CBT

We aim in this study to (1) evaluate the accessibility and effectiveness of MCT and CBT in treating low self-esteem, (2) investigate the patterns of change and the mechanisms of action involved during treatment, and (3) examine the impact of meta-cognitions and neuropsychologial processes in the treatment response and any relapse prevention of low self-esteem.

DETAILED DESCRIPTION:
The association between low self-esteem and psychiatric disorders indicates that low self-esteem is an important transdiagnostic construct. People who report having a low self-esteem seem to experience more mental health problems and a reduction in quality of life.

There have been a few trials considering the effect of Cognitive Behavioural Therapy (CBT) for low self-esteem, however, there are few randomized controlled studies. Recently, Meta Cognitive Therapy (MCT) has been introduced as a new, specific treatment for MDD, showing promising and lasting results. This treatment approach also has proven more effective than CBT for GAD or worry disorder. So far, no study has examined MCT for low self-esteem in a randomized controlled trial.

For the present clinical trial, 20 patients with low self-esteem will be selected and distributed into two treatment conditions. The first group (n=10) will be treated with MCT, whereas the second group (n = 10) will be treated with CBT. The patients will be assessed with different outcome measures at pre-treatment, at the end of treatment, and at six months follow up. In addition, they will also be assessed weekly using various measures.

We aim in this study to (1) evaluate the accessibility and effectiveness of MCT and CBT in treating low self-esteem, (2) investigate the patterns of change and the mechanisms of action involved during treatment, and (3) examine the impact of meta-cognitions and neuropsychologial processes in the treatment response and any relapse prevention of low self-esteem.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to entry in the study.
2. Scores below 15 on the Rosenberg Self-esteem Scale (RSE)
3. 18 years or older.

Exclusion Criteria:

1. Psychosis
2. Bipolar type 1
3. Current suicide intent
4. PTSD
5. Cluster A or cluster B personality disorder
6. Substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self Esteem Scale | Baseline scores each week over two weeks before pre-treatment, pre-treatment, each session each week over 8 weeks , post-treatment (8 weeks), and six months follow up
  The purpose of the 10 item RSE scale is to measure self-esteem.The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem

SECONDARY OUTCOMES:
GAD-7 | Baseline scores each week over two weeks before pre-treatment, pre-treatment, each session each week over 8 weeks, post-treatment (8 weeks) and six months follow up
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day". Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
PHQ-9 | Baseline scores each week over two weeks before pre-treatment, pre-treatment, each session each week over 8 weeks , post-treatment (8 weeks) and six months follow up
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively

OTHER OUTCOMES:
Penn State Worry Questionnaire | Pre-, post-treatment (8 weeks) and six months follow up
  The PSWQ is a 16-item self-report scale designed to measure the trait of worry in adults. Worry is regarded as a dominant feature of generalised anxiety disorder (GAD). The scale measures the excessiveness, generality, and uncontrollable dimensions of worry.cores range from 16 to 80 with higher scores indicative of higher levels of trait worry. Scores can be in the following severity ranges.
  29 or less: Not anxious or a worrier 30-52: Bothered by worries but below clinical range for worry 52-65: Currently have some problems with worry and may benefit from treatment 66 or more: Chronic worrier and in need of treatment to target this problem
Inventory of Interpersonal Problems (IIP-64) | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The Inventory of Interpersonal Problems (IIP) is a self-report instrument that identifies a person's most salient interpersonal difficulties.The questionnaire is divided into two parts. The first part consists of statements about behavior inhibitions commenced 'It's hard for me to…' and the second part includes items that focus on behavioral excesses, 'Things that I do too much…'. The participant responds to the items on a 5-point Likert scale, ranging from 0 = 'Not at all' to 4 = 'Extremely'. Higher scores indicate more interpersonal distress. The items are grouped into eight subscales (with eight items each) corresponding to the octants in the interpersonal circumplex: domineering/controlling (PA), vindictive/self-centered (BC), cold/distant (DE), socially inhibited (FG), non-assertive (HI), overly accommodating (JK), self-sacrificing (LM) and intrusive/needy (NO).
Ruminative Response Scale | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The RRS was developed to more directly and reliably assess rumination that is related to, but not confounded by depression. The 22 items of the RRS measure two aspects of rumination, brooding and reflective pondering.The total score ranges from 22-88, with higher scores indicating increased tendency to ruminate.
Robson Self Concept Questionnaire | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The SCQ is a self-report scale measuring self-esteem. It consists of 30 items (e.g., "I have control over my life," "I feel emotionally mature," "I can like myself even if others don't".It consists of 30 statements to which respondents indicate their level of agreement on a 7-point scale. The typical mean score in control samples being around 140 with a standard deviation of 20.
Metacognitive Questionnaire-30 | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The Metacognitions Questionnaire 30- (MCQ-30) [7] assesses metacognitive beliefs and processes. It comprises five subscales: 'Positive beliefs about worry'; 'Negative beliefs about worry'; 'Cognitive confidence'; 'Need to control thoughts'; and 'Cognitive self-consciousness.Each item is scored on a 4-point scale ranging from 1 ("do not agree") to 4 ("agree very much"). Higher scores reflect more dysfunction with the item in question
BRIEF-A | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The BRIEF-A is composed of 75 items within nine theoretically and empirically derived clinical scales that measure various aspects of executive functioning; Inhibit, Self-Monitor, Plan/Organise, Shift, Initiate,, Task Monitor, Emotional Control, Working Memory, Organisation of Materials. The clinical scales form two broader indexes: Behavioral Regulation (BRI) and Metacognition (MI), and these indexes form the overall summary score, the Global Executive Composite (GEC). The BRIEF- A also includes three validity scales (Negativity, Inconsistency, and Infrequency). All 75 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). Raw scores for each scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning.
CANTAB Intra-Extra Dimensional Set Shift | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The test investigates the processes involved in categorizing stimuli into sets (visual discrimination of shapes vs. lines) and flexible response (shifting of attention) to changes in stimuli.
CANTAB Spatial Working Memory | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The test examines the ability to remember and manipulate visuospatial information
CANTAB Stop Signal Task | Pre-, post-treatment (8 weeks) and six months follow up after treatment
  The test examines the ability to stop a response (response inhibition).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hagen, Professor, Principal Investigator — University of Oslo
Locations (1):
- Department of Psychology, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT06866639/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT06866639/SAP_001.pdf